CLINICAL TRIAL: NCT00139607
Title: A Multicenter, Open Label, Pilot Study To Evaluate Analgesic Activity And Safety Of Parecoxib 40 Mg IV In Patients Undergoing Hemicolectomy, In The Optimal Management Of Acute Post-Operative Pain Of Surgical Patients
Brief Title: Parecoxib In Post Surgery (Hemicolectomy) Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see detailed description for termination reason.
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PARA-0505-079; A3481022
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Colectomy

INTERVENTIONS:
Drug: Paracoxib

SUMMARY:
This is a phase III, multicenter, open label, pilot to evaluate the analgesic efficacy and safety of parecoxib 40 mg IV in the treatment of the pain following hemicolectomy in an optimal management of the surgical patient

DETAILED DESCRIPTION:
The study was terminated prematurely due to recruitment issues on 31 January 2006. Safety concerns did not lead to the decision to terminate this study.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalised for resection of left/right colon;
* preoperative health graded as ASA <3.

Exclusion Criteria:

* patients with any type of metastatic cancer, particularly metastatic colon cancer;
* patients with familial adenomatous polyps (sporadic adenomatous polyps are accepted);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-09; Study Completion 2005-01

PRIMARY OUTCOMES:
Evaluation of efficacy assessments based on pain intensity (VAS) and on Pain relief (PR).

SECONDARY OUTCOMES:
Time between the first administration of parecoxib and the first request of morphine The total amount of morphine in the first 24 hours of treatment and the total amount of morphine given during the entire period of treatment with parecoxib

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Italy (3):
  - Pfizer Investigational Site, Biella
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Siena

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=PARA-0505-079&StudyName=Parecoxib+In+Post+Surgery+%28Hemicolectomy%29+Pain